CLINICAL TRIAL: NCT07070505
Title: Effect of Hand Massage on Physical Restraint Complications
Brief Title: Hand Massage for Physical Restraint
Acronym: Complications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ECE KURT, Lecturer PhD, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Adana City Hospital
Record Dates: First submitted 2025-06-03; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Physical Restraints; Hand Massage

STUDY DESIGN:
Intervention Model Description: Patients in this group will be subjected to routine monitoring as per the hospital procedure every 30 minutes. In addition, one of the patient's wrists that is under restraint will be opened for 5 minutes every 30 minutes and a hand massage will be applied. The open wrist will be restricted again after the 5 minutes are completed. This application will be repeated every 30 minutes until the total restriction period requested by the physician is completed. During the monitoring performed every 30 minutes, the patient's peripheral capillary refill time, skin integrity, skin color, skin temperature and pain will be evaluated and recorded in the Patient Information and Restriction Monitoring Form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients in this group will be subjected to routine monitoring, which is included in the hospital procedure, every 30 minutes. Routine monitoring includes ensuring physical well-being, taking pulse, feeding, giving water, and meeting toilet needs. Records are kept by the nurse regarding these practices. During monitoring every 30 minutes, the patient's peripheral capillary refill time, skin integrity, skin color, skin temperature, and pain will be evaluated and recorded on the Patient Information and Restriction Monitoring Form.
- Experimental group (Experimental): * Before applying hand massage, the individual/patient's hand or arm will be evaluated for thrombus, phlebitis, ecchymosis, hematoma, deterioration in skin integrity and change in skin color in order to determine whether there is a risk.
  * Hand massage application is a massage performed with western technique that includes five basic classical massage manipulations including efflorescence, petrissage, friction, tapotment and vibration.
  * Massage should be performed in a way that creates light pressure on the individual, then the applied pressure should be gradually increased.
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Experimental — * Before applying hand massage, the individual/patient's hand or arm will be evaluated for thrombus, phlebitis, ecchymosis, hematoma, deterioration in skin integrity and change in skin color in order to determine whether there is a risk.
  * Hand massage application is a massage performed with western technique that includes five basic classical massage manipulations including efflorescence, petrissage, friction, tapotment and vibration.
  * Massage should be performed in a way that creates light pressure on the individual, then the applied pressure should be gradually increased.
  Arms: Experimental group

SUMMARY:
In this study, nurses will apply hand massage to patients who are physically restrained. It will be examined whether massage has a positive effect on patients' skin color, blood circulation, skin temperature and pain. Physical restraint will be applied to patients only in the presence of medical indications and with the decision of a physician.

Research question: Does hand massage applied to patients in physical restraint have an effect on preventing complications related to restraint?

DETAILED DESCRIPTION:
There are 2 groups in the study: experimental and control. Patients in the control group will be subjected to the hospital's routine physical restraint practices and will not receive hand massage.

ELIGIBILITY:
Inclusion Criteria:

* Both physical and chemical restraint must be applied, a written request for restraint must be given by the physician, both upper extremities must be restrained, and verbal permission must be obtained from the relatives.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
During the 30. 60th. 90. 120. minutes follow-up, the patient's peripheral capillary refill time, skin integrity, skin color, skin temperature and pain will be evaluated. | for 2 hours
  Peripheral capillary refill time
  ( 0-2 sec : + ) ( >2 sec : ++ ) Skin integrity + yes
  - no
  If yes, specify:
  * abrasion
  * irritation
  * laceration Specify skin color
  * Pale/white
  * red
  * bruised
  * pink Skin temperature
  Compared to unrestricted area
  * warmer
  * colder
  * no difference Pain (0-10 points) Ask the patient about the restricted area
    0: I have no pain
    10: Unbearable pain 30th min 60th min 90th min 120th min

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Ekrem Tok Mental Health Hospital, Adana, Turkey (Türkiye)